CLINICAL TRIAL: NCT00203255
Title: An Open-Label, Pilot Study Examining the Use of Soy Isoflavones in the Prevention of Menstrually-Associated Migraine
Brief Title: Clinical Study Examining Use of an Over-the-Counter Supplement for the Prevention of Menstrually-Associated Migraine Headache
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Thomas Jefferson University (Other)
Collaborators: Johnson & Johnson (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None
Other Study IDs: SDS/SOY/02
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2009-01-23 (Estimated); Status verified 2009-01

CONDITIONS: Migraine Headache
Keywords: Menstrually-Associated Migraine
MeSH Terms: conditions — Migraine Disorders | interventions — Soybean Proteins

INTERVENTIONS:
Drug: Soy Isoflavones

SUMMARY:
The purpose of this trial is to study the use of soy isoflavones in the prevention of menstrually-associated migraines. Additionally, this trial may provide insight into the menstrual cycle and menstrually-related headaches in women. With this information, we may be able to change current treatment methods or even develop new methods in order to advance current approaches in the treatment of menstrual migraine.

DETAILED DESCRIPTION:
Many women have increased headache attacks at the time of their period (menses). The migraines experienced around the menstrual cycle are most often associated with premenstrual complaints such as nausea, backache and breast tenderness. The condition of hormone-related headache (i.e. menstrual migraine) is unclear.

Soy isoflavones have been used to alleviate the symptoms of menopause. They contain natural estrogens (female hormones). Since menstrual migraine is thought to be associated with the withdrawal of estrogen, or the natural fall of estrogen levels, the use of this natural source of estrogen may be helpful in the prevention of menstrually-associated migraine.

ELIGIBILITY:
Inclusion Criteria:

•Subjects who have experienced regular menstrual cycles for the past 6 months (every 21 to 35 days) •Subjects who have a history of migraine with or without aura that meets IHS criteria for at least 6 months preceding the study. •Subjects who have headaches associated with menstruation, either pre-menstrually or menstrually (defined as from day -3 through the cessation of menstrual flow) at least 75% of the time (3 out of the past 4 months). •Subjects must experience a menstrually-associated migraine during the baseline month, as defined above. •Subjects must be able to accurately predict onset on menses (within 2 days). This will be confirmed during the baseline month. •Subjects who have been on stable headache preventive medications for the 3 months prior to screening. •Subject has negative urine pregnancy test prior to study entry, and is using or agrees to use for the duration of participation a medically acceptable form of contraception (as determined by investigator), if female of child-bearing potential •Subject is able to understand and comply with all study requirements •Subject provides written informed consent prior to any screening procedures being conducted

Exclusion Criteria:

* Subjects who are breastfeeding, pregnant or planning to become pregnant within the next 4 months. •Subjects who are currently on or have been on within three months prior to screening; hormonal contraceptives (oral, injection, or implants), hormone replacement therapy or any other hormone therapy including natural supplements. •Subjects who, in the investigators opinion, have a history or have evidence of a medical or psychiatric condition that would expose them to an increased risk of a significant adverse event or would interfere with the assessments of efficacy and tolerability during this trial •Subjects who experience greater than 15 headache days per month •Subjects who have an allergy to soy or soy based products. •Subjects with a history of significant drug or alcohol abuse within the past year
* Subjects who have participated in an investigational drug trial in the 30 days prior to the screening visit •Subjects who have breast cancer or who have a history of breast cancer.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25
Dates: Start 2003-05; Study Completion 2005-03

PRIMARY OUTCOMES:
To compare headache outcome measures between baseline and soy treatment periods. Headache outcome measures include frequency and duration of menstrually-associated migraine (MAM), as well as presence or absence of associated symptoms

SECONDARY OUTCOMES:
Duration of MAM headaches
Maximum headache intensity
Incidence of MAM headache associated symptoms
Duration of MAM headache associated symptoms
Maximum functional impairment score during MAM headache
Incidence of use of rescue medication for the treatment of a MAM attack
Patient satisfaction score at the end of each treatment period
Describe headaches associated with menstruation
Describe the association of headache to premenstrual symptoms.
Explore premonitory symptoms in the menstrual migraine population
Compare questionnaire data collected at screening visit to questionnaire data collected at termination visit.
Assess electronic diary effectiveness in capturing diary information in this population

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D. Silberstein, M.D., Principal Investigator — Thomas Jefferson University, Jefferson Headache Center
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States